CLINICAL TRIAL: NCT04773366
Title: A Prospective Institutional Study for the Treatment of Children With Newly Diagnosed Langerhans Cell Histiocytosis Using a Cytarabine Contained Protocol
Brief Title: A Prospective Study for the Treatment of Children With Newly Diagnosed LCH Using a Cytarabine Contained Protocol
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCMC-LCH-2018
Record Dates: First submitted 2021-02-18; First posted 2021-02-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Langerhans cell histiocytosis; pediatric patients; cytarabine; treatment outcome
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Hyperthermia, Induced

STUDY DESIGN:
Intervention Model Description: All enrolled patients are stratified into 4 risk groups. Patients in each risk group are assigned to one treatment regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Multisystem patients (≥2 organs/systems) with involvement of one or more "Risk" organs, i.e. hematopoietic system, liver or spleen.
  All patients in this group receive an initial therapy (Week 1~6) followed by a consolidation continuation therapy (Week 7~22) and maintenance continuation therapy (Week 25~52).
  Interventions: Drug: Prednisone+Cytarabine+vincristine; Drug: Prednisone+Cytarabine+vincristine+Mercaptopurine
- Group 2 (Experimental): Multisystem patients, but without involvement of "Risk" organs.
  All patients in this group receive an initial therapy (Week 1~6) followed by continuation therapy (Week 7~52).
  Interventions: Drug: Prednisone+Cytarabine+vincristine; Drug: Prednisone+vincristine+Mercaptopurine
- Group 3 (Experimental): Includes patients with single system, multifocal or with single system, unifocal and special site (Isolated lesion of special site) or with single system, unifocal and CNS risk or with single system, unifocal i.e. thyroid, lung, thymus, hypothalamic-pituitary or with single system, unifocal and other functionally critical anatomical sites.
  All patients in this group receive an initial therapy (Week 1~6) followed by continuation therapy (Week 7~52).
  Interventions: Drug: Prednisone+vincristine
- Group 4 (Experimental): Patients with single system, unifocal i.e. bone, skin or lymph node (not the draining lymph node of another LCH lesion).
  All patients in this group enter into observation after local therapy. Chemotherapy only apply to patients with disease reactivation during observation.
  Interventions: Other: Local therapy

INTERVENTIONS:
Drug: Prednisone+Cytarabine+vincristine — Group 1 initial treatment (W1~W6). Prednisone 40mg/m2×4w, taper 2w; Vincristine 1.5mg/m2 iv d1 of w1,2,3,4,5,6; Cytarabine 100mg/m2 iv/IH d1-4 q2w (w1,3,5)
  Arms: Group 1
Drug: Prednisone+Cytarabine+vincristine+Mercaptopurine — Group 1 Consolidation continuation treatment (W7~W22) . Prednisone 40mg/m2 d1-5 q3w (w7,10,13,16,19,22); VCR 1.5/m2 iv d1 q3w (w7,10,13,16,19,22); Cytarabine 100mg/m2 iv/IH d1-4 q3w (w7,10,13,16,19,22); 6-MP 50mg/m2/d,po,qn
  Arms: Group 1
Drug: Prednisone+Cytarabine+vincristine+Mercaptopurine — Group 1 Maintenance continuation treatment (W25~52) . Prednisone 40mg/m2 d1-5 q3w; Vincristine 1.5/m2 iv d1 q3w; Cytarabine 100mg/m2 iv/IH d1-4 q6w ×3 times (w25,31,37); 6-MP 50mg/m2/d,po,qn
  Arms: Group 1
Drug: Prednisone+Cytarabine+vincristine — Group 2 Initial treatment (W1~W6) . Prednisone 40mg/m2×4w, taper 2w; Vincristine 1.5mg/m2 iv d1 of w1,2,3,4,5,6; Cytarabine 100mg/m2 iv/IH d1-4 q2w (w1,3,5)
  Arms: Group 2
Drug: Prednisone+vincristine+Mercaptopurine — Group 2 continuation treatment (W7~W52) . Prednisone 40mg/m2 d1-5 q3w; VCR 1.5/m2 iv d1 q3w; 6-MP 50mg/m2/d,po,qn
  Arms: Group 2
Drug: Prednisone+vincristine — Group 3 Initial treatment (W1~W6) . Prednisone 40mg/m2×4w, taper 2w; Vincristine 1.5mg/m2 iv d1 of w1,2,3,4,5,6
  Arms: Group 3
Drug: Prednisone+vincristine — . Group 3 Continuation treatment (W7~W52)Prednisone 40mg/m2 d1-5 q3w; Vincristine 1.5/m2 iv d1 q3w
  Arms: Group 3
Other: Local therapy — Local therapy/wait and see. Group 4
  Arms: Group 4

SUMMARY:
From January 2010 to December 2014, 150 children with MS-LCH were treated in our hospital following a LCH II (Arm B) based protocol. Treatment was based on a modification of the LCH-II (Arm B) based protocol. However, the continuation treatment was extended to 56 weeks and etoposide was omitted from the continuation treatment.

For the 59 patients with RO involvement (RO+) (the lungs are not considered a RO in the current study), the rapid response rate (week 6) was 61.0% and the 3-year overall survival (OS) 73.4±5.9%. Rapid responders had a better 3-year survival rate than poor responders (90.9±5.0% vs. 45.7±11.0%, P<0.001). The 3-year OS in the current study is 10~20% lower than the rates reported by Gadner et al. and Morimoto et al.. We have not yet adopted effective salvage therapies for RO+ patients with recurrent disease. During the time of this study, cladribine was unavailable. Second-line therapy for non-responders or patients with disease reactivation was individualized treatment based on the physician's experience. An effective salvage therapy is essential for this high-risk group.

For 91without RO involvement (RO-), 78 patients (85.7%) were rapid responders at week 6. The 3-year cumulative reactivation rate was 10.7% for RO- patients. No death occurred in this subgroup, with a 3-year OS of 100% in RO- patients. Compared to the LCH II and LCH III trials, the current study had a more intensive initial treatment regimen for RO- patients. However, the addition of etoposide to prednisone and vincristine in the initial therapy did not increase the 6-week response rate for RO- patients (85.7% in this study compared to 83% in the LCH II study and 86% in the LCH III study). Surprisingly, with a relatively intense initial treatment, a relatively low 3-year cumulative reactivation rate was observed in RO- patients in the current study. This result suggests that the initial treatment intensity and duration of continuation therapy both impact disease reactivation. The intensity of induction can affect the degree of disease resolution. Insufficient treatment intensity might lead to late relapse. Similarity to that observed has been in other childhood hematological malignancies. This finding deserves to be tested in prospective clinical trials with long-term follow-up. Cytarabine has been applied for patients with LCH but has never been evaluated in our hospital prospectively. In this study, we administer a cytarabine contained protocol to patients with multisystem involvement with or without risk organs involvement. The treatment results will be compared with our historical studies.

DETAILED DESCRIPTION:
All patients with de novo pathological confirmed LCH enrolled in this study will be classified into 4 groups. Group 1: Multisystem patients (≥2 organs/systems) with involvement of one or more "Risk" organs" (hematopoietic system, liver or spleen);Group 2:Multisystem patients, but without involvement of "Risk" organs; Group 3: Single system, Multifocal+ Single system, unifocal and special site@ (Isolated lesion of special site)+ Single system, unifocal and CNS risk+Single system, unifocal i.e. thyroid, lung, thymus, hypothalamic-pituitary+Single system, unifocal and other functionally critical anatomical sites; Group 4: Single system, unifocal i.e. bone, skin or lymph node (not the draining lymph node of another LCH lesion). For patients in Group 1, a 6-week initial treatment, a 16-week consolidation continuation treatment and a 26-week maintenance continuation treatment containing cytarabine is applied. For patients in Group 2, a 6-week initial treatment containing cytarabine and a 46-week continuation treatment (without cytarabine) is applied. For patients in Group 3,a 6-week initial treatment and a 46-week continuation treatment (without cytarabine) is applied. For patients in Group 4, only local therapy followed by wait-and-see strategy is applied.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 18 years
2. Newly diagnosed LCH：Morphologic identification of the characteristic LCH cells, positive staining of the lesional cells with CD1α and/or Langerin
3. No congenital immunodeficiency, HIV infection, or prior organ transplant
4. No previous chemotherapy/target therapy/radiation, if any steroid applied, total prior steroids dosage < prednisone 280 mg/m2

Exclusion Criteria:

* Patients have overwhelming infection, and a life expectancy of < 2 weeks

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of responders after initial treatment for patients with risk organ involvement | Evaluation at week 6 or 12
  Rate of responders after initial treatment and consolidation continuation treatment. A good response is defined as complete resolution (no evidence of active disease) in risk organs.
Reactivation rate for all patients | Up to 5 years
  Reactivation is defined as progression or relapse in any organ or system after disease complete resolution (no evidence of active disease).

SECONDARY OUTCOMES:
Overall survival for patients with risk organ involvement | Up to 5 years
  Overall survival is measured using the Kaplan-Meier method. From the day of diagnosis to death for any reason or to the date of the last follow-up contact.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

REFERENCES:
- [Background] Simko SJ, McClain KL, Allen CE. Up-front therapy for LCH: is it time to test an alternative to vinblastine/prednisone? Br J Haematol. 2015 Apr;169(2):299-301. doi: 10.1111/bjh.13208. Epub 2014 Nov 16. No abstract available. PMID 25400231
- [Background] Gadner H, Grois N, Potschger U, Minkov M, Arico M, Braier J, Broadbent V, Donadieu J, Henter JI, McCarter R, Ladisch S; Histiocyte Society. Improved outcome in multisystem Langerhans cell histiocytosis is associated with therapy intensification. Blood. 2008 Mar 1;111(5):2556-62. doi: 10.1182/blood-2007-08-106211. Epub 2007 Dec 18. PMID 18089850
- [Background] Gadner H, Grois N, Arico M, Broadbent V, Ceci A, Jakobson A, Komp D, Michaelis J, Nicholson S, Potschger U, Pritchard J, Ladisch S; Histiocyte Society. A randomized trial of treatment for multisystem Langerhans' cell histiocytosis. J Pediatr. 2001 May;138(5):728-34. doi: 10.1067/mpd.2001.111331. PMID 11343051
- [Background] Egeler RM, de Kraker J, Voute PA. Cytosine-arabinoside, vincristine, and prednisolone in the treatment of children with disseminated Langerhans cell histiocytosis with organ dysfunction: experience at a single institution. Med Pediatr Oncol. 1993;21(4):265-70. doi: 10.1002/mpo.2950210406. PMID 8469221
- [Background] Weitzman S, Braier J, Donadieu J, Egeler RM, Grois N, Ladisch S, Potschger U, Webb D, Whitlock J, Arceci RJ. 2'-Chlorodeoxyadenosine (2-CdA) as salvage therapy for Langerhans cell histiocytosis (LCH). results of the LCH-S-98 protocol of the Histiocyte Society. Pediatr Blood Cancer. 2009 Dec 15;53(7):1271-6. doi: 10.1002/pbc.22229. PMID 19731321
- [Background] Donadieu J, Bernard F, van Noesel M, Barkaoui M, Bardet O, Mura R, Arico M, Piguet C, Gandemer V, Armari Alla C, Clausen N, Jeziorski E, Lambilliote A, Weitzman S, Henter JI, Van Den Bos C; Salvage Group of the Histiocyte Society. Cladribine and cytarabine in refractory multisystem Langerhans cell histiocytosis: results of an international phase 2 study. Blood. 2015 Sep 17;126(12):1415-23. doi: 10.1182/blood-2015-03-635151. Epub 2015 Jul 20. PMID 26194764
- [Background] Braier J, Rosso D, Pollono D, Rey G, Lagomarsino E, Latella A, Zubizarreta P. Symptomatic bone langerhans cell histiocytosis treated at diagnosis or after reactivation with indomethacin alone. J Pediatr Hematol Oncol. 2014 Jul;36(5):e280-4. doi: 10.1097/MPH.0000000000000165001. PMID 24977402
- [Background] Heritier S, Jehanne M, Leverger G, Emile JF, Alvarez JC, Haroche J, Donadieu J. Vemurafenib Use in an Infant for High-Risk Langerhans Cell Histiocytosis. JAMA Oncol. 2015 Sep;1(6):836-8. doi: 10.1001/jamaoncol.2015.0736. No abstract available. PMID 26180941
- [Result] Gao YJ, Su M, Tang JY, Pan C, Chen J. Treatment Outcome of Children With Multisystem Langerhans Cell Histiocytosis: The Experience of a Single Children's Hospital in Shanghai, China. J Pediatr Hematol Oncol. 2018 Jan;40(1):e9-e12. doi: 10.1097/MPH.0000000000001016. PMID 29200145
- [Result] Su M, Gao YJ, Pan C, Chen J, Tang JY. Outcome of children with Langerhans cell histiocytosis and single-system involvement: A retrospective study at a single center in Shanghai, China. Pediatr Hematol Oncol. 2018 Oct-Nov;35(7-8):385-392. doi: 10.1080/08880018.2018.1545814. Epub 2019 Jan 29. PMID 30693828
- [Result] Gadner H, Minkov M, Grois N, Potschger U, Thiem E, Arico M, Astigarraga I, Braier J, Donadieu J, Henter JI, Janka-Schaub G, McClain KL, Weitzman S, Windebank K, Ladisch S; Histiocyte Society. Therapy prolongation improves outcome in multisystem Langerhans cell histiocytosis. Blood. 2013 Jun 20;121(25):5006-14. doi: 10.1182/blood-2012-09-455774. Epub 2013 Apr 15. PMID 23589673